CLINICAL TRIAL: NCT06436456
Title: The Feasibility, Acceptability and Preliminary Effectiveness of an Internet-based Intervention for Diabetes Distress in Patients With Type 1 Diabetes
Brief Title: Use of an Online Intervention for the Treatment of Diabetes Distress in Patients With Type 1-Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Center for Digital Psykiatri (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22/57849
Record Dates: First submitted 2024-05-03; First posted 2024-05-31 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Distress
Keywords: Diabetes Mellitus, Type 1; Diabetes distress; Online intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: 1. Online psychological intervention
  2. Individual psychological intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online psychological intervention (Experimental): Online psychological intervention with written support from a psychologist
  Interventions: Behavioral: Online psychological intervention
- Individual psychological intervention (Active Comparator): Individual therapy sessions with a psychologist
  Interventions: Behavioral: Individual psychological intervention

INTERVENTIONS:
Behavioral: Online psychological intervention — The online intervention constitutes a psychological intervention rooted in therapeutic principals of Acceptance and Commitment Therapy (ACT) and Cognitive Behavioral Therapy (CBT). Comprising 7 obligatory modules and 4 optional modules, the intervention is facilitated through an online platform, offering a text-based self-help program. Patients receive written guidance from a psychologist at Steno Diabetes Center Odense (SDCO). While undergoing intervention, patients have the option to seek clarification or assistance from the psychologist if encountered with queries or difficulties. It is anticipated that patients will progress through approximately one module per week. Following completion of the intervention, patients retain access to the online intervention for a duration of 3 months.
  Arms: Online psychological intervention
Behavioral: Individual psychological intervention — In the individual intervention, patients undergo personalized therapy administered by the assigned psychologist from SDCO. This treatment approach is grounded in the principles of Acceptance and Commitment Therapy (ACT) and Cognitive Behavioral Therapy (CBT). Delivery of treatment can occur through various modalities, including telephone, video conferencing, or in-person sessions, tailored to accommodate the preferences and requirements of the patient. A maximum of 10 treatment sessions are available for each patient.
  Arms: Individual psychological intervention

SUMMARY:
This study will investigate whether an online intervention can be helpful in reducing diabetes distress in people with type 1 diabetes and elevated diabetes distress, compared to individual counselling sessions (online, phone-based or face-to-face, depending on the preference of the person with type 1 diabetes). Half of the participants will receive the online intervention, while the other half will receive individual counseling sessions with a psychologist.

Objectives: The main aim of this study is to investigate if the online intervention is feasible and liked by people with type 1 diabetes and diabetes distress, in comparison with individual counselling sessions.

Hypotheses: The investigators predict that both interventions will be feasible to use, shown by how many people join, stay engaged, and complete the interventions. The investigators also think that people will find both interventions acceptable, as shown by the positive feedback given in interviews after they finish.

DETAILED DESCRIPTION:
Individuals with diabetes are primarily responsible for managing their disease. Therefore, their ability to effectively self-treat their diabetes is critical for their prognosis. These significant treatment responsibilities place considerable demands on individual patients. These demands can lead to high levels of diabetes distress. Diabetes distress encompasses the emotional distress arising from the constant self-care burden that is required to self-manage diabetes, but also feelings of insufficient support and understanding from others, and challenges in communication with healthcare professionals. Diabetes distress is prevalent among individuals with diabetes. International research indicates that approximately 20-25% of individuals with diabetes experience high levels of diabetes distress. Studies exploring the impact of diabetes distress on diabetes management reveal that significant diabetes distress not only diminishes overall well-being but also correlates with suboptimal self-management of diabetes. This includes insufficient physical activity, unhealthy dietary choices, reduced medication adherence, infrequent blood glucose monitoring, and elevated HbA1c levels.

At Steno Diabetes Center Odense (SDCO), there are provisions for individual psychological intervention aimed at patients facing psychological challenges associated with their diabetes. However, due to resource constraints, priority is given to those patients experiencing the most severe impact.

As part of a new initiative at SDCO, Patient-Reported Outcome (PRO) data has been incorporated alongside diabetes same-day micro- and macrovascular complication screening, which includes an assessment of mental well-being (i.e. diabetes distress). These assessments will contribute to higher recognition rates of elevated diabetes distress, thereby exacerbating the strain on already limited resources available for individual psychological intervention. Moreover, not all patients may have the requisite time, necessity, or opportunity to partake in such individual intervention.

In order to expand existing psychological services at SDCO in an affordable way, an online psychological intervention needs to be developed. The objective of the online psychological intervention is to cater to a larger group of people with type 1 diabetes, who can autonomously engage with evidence-based components of the intervention, thereby averting the progression of patients' diabetes distress towards adverse or pathological conditions, such as anxiety or depression. Studies indicate that therapist-supported online therapy yields comparable efficacy to traditional face-to-face therapy. Additionally, online therapy offers the benefit of flexibility, allowing patients to engage with the intervention at their convenience, thereby obviating the need for patients to take time away from their professional commitments to attend sessions with a psychologist.

Aims:

The primary aim of this study is to evaluate the feasibility and acceptability of an online intervention with written support for patients with type 1-diabetes and elevated diabetes distress, comparing this with an individual intervention by a psychologist (online, phone-based or face-to-face, depending on the preference of the person with type 1 diabetes). Following the intervention, qualitative data will be collected through interviews conducted with both patients and clinical staff to assess this aim. Also metadata from the platform of the online intervention will be collected to evaluate this aim.

A secondary aim is to explore the efficacy of the interventions to improve different domains of diabetes-stress. This secondary aim will be evaluated through survey data.

Further aims are to explore whether both interventions impact diabetes-related quality of life, acceptance of diabetes, patient engagement in healthcare, negative effects of the intervention, useability of the intervention and glucometrics (e.g. estimated HbA1c, time in range (TIR), time above range (TAR), time below range (TBR)).

Hypotheses:

Primary aim hypotheses: It is hypothesized that both interventions will show high feasibility and acceptability, demonstrated by acceptable recruitment strategies, high rates of retention and high completion of modules/sessions. It is expected though, that the dropout rates will be higher in the online intervention group. It is also hypothesized that both interventions are acceptable, as demonstrated by satisfactory feedback obtained through post-intervention interviews.

Secondary aim hypotheses. It is hypothesized that in both interventions there will be a significant reduction in participants' diabetes distress from pre-intervention to post-intervention, and from pre-intervention to 3-months follow-up.

Further, it is also hypothesized that the interventions will yield positive changes in diabetes-related quality of life, acceptance of diabetes, and patient engagement in healthcare. It is further hypothesized that the interventions has no negative effect on the patients, and that the patients find the interventions useful. Glucometrics are included as a secondary outcome but as the interventions does not target this, the investigators hypothesize no changes in these measures will be found.

Recruitment and procedure:

Participants for the study will be recruited at Steno Diabetes Center Odense (SDCO) in Denmark. Patients with a total score on the questionnaire Problem Areas in Diabetes (PAID5) of ≥ 8 will receive information about the study. If interested in participating, they can contact the study leader to receive more information about the study and schedule a screening appointment with a study psychologist.

During the screening appointment, the patient will have further opportunity to learn more about the study and ask questions. If they wish to participate, they will receive a consent form to sign. Subsequently, the patient will receive a questionnaire including an extended measure of diabetes distress i.e. The Diabetes Distress Scale for type 1-diabetes (DDS-type1). In the screening appointment, the inclusion and exclusion criteria will be evaluated. If the psychologist deems the patient suitable for participation, the patient will be randomized to either receive an online psychological intervention or an individual psychological intervention with 20 patients in each arm.

Following the conclusion of the intervention and during the 3-month follow-up period, participants will be administered a questionnaire.

Subsequent to the feasibility study, semi-structured interviews will be conducted with approx. 12 patients, 2-3 psychologists, and possibly further clinical staff. These interviews will explore aspects related to screening procedures, recruitment strategies, and the acceptance of the online psychological intervention.

The online intervention will subsequently be evaluated using a mini Model for Assessment of Telemedicine (MAST), where the following domains will be assessed:

* Health problems and technology characteristics
* Patient safety
* Clinical effectiveness
* Patient assessment
* Economic aspects
* Organizational aspects
* Sociocultural, ethical, and legal aspects.

ELIGIBILITY:
Inclusion Criteria:

* A total score or a score on one of the subscales of the Diabetes Distress Scale for type 1 diabetes which is 2 or above.
* Diagnosed with type 1-diabetes ≥ 12 months ago.
* Age ≥ 30 years.
* Receiving treatment at SDCO.
* Proficiency in Danish and basic IT skills.

Exclusion Criteria:

* Psychiatric diagnosis that may compromise participation in the intervention e.g. psychosis, schizophrenia, substance or alcohol abuse.
* Cognitive impairments that may compromise participation in the intervention e.g. dementia, Alzheimer's, brain injury.
* Complex issues best suited for individual treatment as assessed by the clinical psychologist.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of eligible patients who agree to participate in the interventions throughout the study period | Throughout the duration of the study approx. 12 months
  The number of eligible patients who agree to participate in the interventions
The completion rates of survey measures at pre- and post-intervention and at three months follow-up | Immediately before enrollment in the intervention, immediately after the intervention and three months after the intervention
  The number of patients completing the survey measures at pre- and post-intervention as well as at three months follow-up
Characteristics of patients receiving the interventions and those who drop out assessed through survey data. | Throughout study participation, an average of 6 months
  Patient characteristics assessed through survey data
Acceptability of the online intervention expressed by patients | After completion of the intervention, an average of 3-12 months
  Will be assess by expressions of patients through qualitative semi structured interviews
Acceptability of the online intervention expressed by participating clinical staff | Obtained after study completion approx.12 months
  Will be assess by expressions of participating clinical staff through qualitative semi structured interviews
Number of log ins on the platform | Obtained after completion of the online intervention, an average of 3-6 months
  The number of log ins on the platform by patients in the online intervention
Time points of log ins on the platform | Obtained after completion of the online intervention, an average of 3-6 months
  The time points of log ins to the platform by patients in the online intervention during their access to the platform
Numbers of hours spend on the platform | Obtained after completion of the online intervention, an average of 3-6 months
  The number of hours the patients in the online intervention spend on the platform during their access to the platform
Numbers of modules completed in the online intervention | Obtained after completion of the online intervention, an average of 3-6 months
  The number of modules completed by the patients in the online intervention
Number of messages sent between patients and psychologist | Obtained after completion of the online intervention, an average of 3-6 months
  The number of messages sent between the patients in the online intervention and their psychologist

SECONDARY OUTCOMES:
Diabetes Distress Scale for type 1 diabetes (T1 DDS) | Immediately before enrollment in the intervention, immediately after the intervention and three months after the intervention
  The T1 DDS measures diabetes distress. The scale consists of 28 items with each item with 6 answer categories ranging from 1 'Not a problem' to 6 'A serious problem'. A total score is calculated by adding all the items together and diving the number by 28. A score between 2,0 and 2,99 indicated moderate diabetes distress and a score of ≥ 3 indicate high levels of diabetes distress
Acceptance & Action Diabetes Questionnaire (AADQ-6) | Immediately before enrollment in the intervention, immediately after the intervention and three months after the intervention
  The AADQ-6 measures diabetes acceptance through 6 items with scores ranging from 1 'Never' to 5 'Almost always'.The scores range from 6-30 with higher values indicate greater non-acceptance
The Patient Activation Measure (PAM) | Immediately before enrollment in the intervention, immediately after the intervention and three months after the intervention
  The PAM assesses patient engagement in healthcare. Three key domains are assessed to understand a person's self-management ability: Knowledge, Skills, Confidence. The scale has 13 items with four answer categories from 'Highly agree' to 'Highly disagree' and a 'Do not know' category. The scores are calculated through an excel spreadsheet created by InsigniaHealth and range from 0-100 with higher scores indicating higher patient activation.
The DAWN (Diabetes Attitudes, Wishes and Needs study) Impact of Diabetes Profile (DIDP) | Immediately before enrollment in the intervention, immediately after the intervention and three months after the intervention
  The DIPD measures diabetes-related quality of life. There scale has 6 items assessing how diabetes affect the following areas (physical health, mental health, relationships, leisure activities, work or studies, financial situation), and two optional items (ability to eat what one wants and overall happiness). Each item can be evaluated using a 7-point scale, where 1 indicates 'A very positive impact', 4 indicates 'No impact', and 7 indicates 'A very negative impact'. Additionally, there is a "not applicable" (N/A) response option available for each item. A higher score indicates lower diabetes-related quality of life.
Negative Effect Questionnaire (NEQ) | Immediately after the intervention
  The NEQ measures negative effects in psychological treatments. It consists of 20 items. First, participants indicate whether specific items occurred during treatment with a binary response (1 for 'Yes', 0 for 'No'). Second, they rate the severity of negative effects on a four-point Likert scale, ranging from 0 'Not at all' to 4 'Extremely'. Third, respondents attribute negative effects to either 1 'The treatment received' or 0 'Other circumstances'. The sum of these items provides a frequency measure of the negative effects experienced by respondents, categorized by treatment or other circumstances.
System Usability Scale (SUS) | Immediately after the online intervention
  The SUS generates a singular numerical value representing a composite measure of the overall usability of the system being studied. Each item's contribution ranges from 1 'Strongly disagree' to 5 'Strongly agree'. For items 1, 3, 5, 7, and 9, the contribution equals the position on the scale minus 1. Conversely, for items 2, 4, 6, 8, and 10, the contribution equals 5 minus the scale position. After summing the scores, the total is multiplied by 2.5 to acquire the overall SUS value. SUS scores range from 0 to 100.
Estimated HbA1c | Pre-intervention (approx. one month before the intervention) and after the intervention (approx. one month after the intervention)
  HbA1c is calculated based on data from the patients' sensor. The unit for reporting HbA1c concentration is mmol/mol
Time in range (TIR) is the percentage of time the blood glucose levels in the recommended target range | Pre-intervention (approx. one month before the intervention) and after the intervention (approx. one month after the intervention)
  TIR is calculated based on data from the patients' sensor - set at the range 3.9-10.0 mmol/L
Time below range (TBR) is the percentage of time the blood glucose levels is below the recommended target range | Pre-intervention (approx. one month before the intervention) and after the intervention (approx. one month after the intervention)
  TBR is calculated based on data from the patients' sensor i.e. below 3.9 mmol/L
Time above range (TAR) is the percentage of time the blood glucose levels is above the recommended target range | Pre-intervention (approx. one month before the intervention) and after the intervention (approx. one month after the intervention)
  TAR is calculated based on data from the patients' sensor i.e. above 10.0 mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Odense, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No